#### STATISTICAL ANALYSIS PLAN

A Multicenter, Randomized, Double-blind,
Vehicle-controlled, Parallel-group Trial to Assess the Safety and
Efficacy of 0.3% and 1% OPA-15406 Ointments When
Administered for 4 Weeks in Pediatric Patients With
Atopic Dermatitis

NCT Number: 03018691

PRT NO. : 271-102-00002

PRT Version Date: 9 Aug 2017 (Version 1)

# A Multicenter, Randomized, Double-blind, Vehicle-controlled, Parallel-group Trial to Assess the Safety and Efficacy of 0.3% and 1% OPA-15406 Ointments When Administered for 4 Weeks in Pediatric Patients With

Atopic Dermatitis

Phase 2

# STATISTICAL ANALYSIS PLAN

for

Protocol No. 271-102-00002

(Translated Version)

#### Confidential

Otsuka Pharmaceutical Co., Ltd

Version 1: 9 Aug 2017

Date of Translation: 28 Nov 2017

# **Table of Contents**

| Tab | Γable of Contents | |
|---|---|---|
| List | of Abbreviations and Definition of Terms | 5 |
| 1 | Introduction | 6 |
| 2 | Trial Objectives | 6 |
| 3 | Trial Design | |
| 4 | Implementation of Planned Analyses | |
| 5 | Statistical Analysis Sets | |
| 5.1 | Definitions of Analysis Sets | |
| 6 | Considerations for Data Analysis | |
| 6.1 | Software | |
| 6.2 | Dictionaries | |
| 6.3 | Data Conversion and Calculation | 9 |
| 6.4 | Study Week Windows | 11 |
| 6.5 | Handling of Missing Values | 12 |
| 6.6 | Significance Level and Confidence Coefficient | 12 |
| 7 | Disposition of Subjects | 13 |
| 7.1 | Disposition of Subjects | 13 |
| 7.2 | Statistical Analysis Sets | 13 |
| 7.3 | Protocol Deviations | 13 |
| 8 | Description of Analysis Datasets | 13 |
| 8.1 | Demographics and Baseline Characteristics | 13 |
| 8.2 | Medical History/Complications | 14 |
| 8.3 | Prior and Concomitant Medications | 14 |
| 8.4 | Concomitant Therapies | 14 |
| 9 | Safety Analysis | 14 |
| 9.1 | Primary Endpoint | 14 |
| 9.2 | Exposure to the IMP (Number of Subjects, Duration, and Doses) | 14 |
| 9.3 | Adverse Events | 15 |
| 9.4 | Potentially Drug-related TEAEs | 15 |

#### Protocol 271-102-00002

| 9.5 | Clinical Laboratory Tests | 15 |
|---|---|---|
| 9.6 | Vital Signs (Including Body Weight) | 16 |
| 9.7 | Electrocardiogram (12-Lead ECG) | 16 |
| 10 | Efficacy Analyses | 17 |
| 10.1 | Secondary Endpoints | 17 |
| 10.2 | Other Efficacy Endpoints | 21 |
| 10.3 | Adjustments for Covariates | 22 |
| 10.4 | Subgroup Analysis | 22 |
| 11 | Pharmacokinetic Analyses | 22 |
| 11.1 | Pharmacokinetics Analysis Set | 22 |
| 11.2 | Pharmacokinetic Endpoints | 22 |
| 11.3 | Method of Calculation of Pharmacokinetic Endpoints | 22 |
| 11.4 | Method of Display | 23 |
| 11.5 | Handling of Values | 23 |
| 12 | Rationale for Target Number of Subjects | 24 |
| 12.1 | Target Number of Subjects | 24 |
| 12.2 | Rationale for the Number of Subjects | 24 |
| 13 | Changes From Analysis Planned in the Protocol | 24 |
| 13.1 | Changes From the Efficacy Analyses Planned in the Protocol | 24 |
| 13.2 | Changes From the Pharmacokinetic Analyses Planned in the Protocol | 24 |
| 14 | References | 25 |
| 15 | Revision History | 26 |
| 16 | Appendix | 27 |
| 16.1 | Criteria for Potentially Clinically Significant | |
| 16.2 | Table of Contents | 28 |

# **List of Abbreviations and Definition of Terms**

# **List of Abbreviations**

| <b>Abbreviation Expansion</b> | |
|---|---|
| AD | Atopic Dermatitis |
| BSA | Body Surface Area |
| EASI | Eczema Area and Severity Index |
| IGA | Investigator's Global Assessment |
| IMP | Investigational Medicinal Product |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed Model Repeated Measures |
| OC | Observed Cases |
| POEM | Patient-Oriented Eczema Measure |
| QTcB | QT interval as correlated by Bazett's formula |
| QTcF | QT interval as correlated by Fridericia's formula |
| SS | Safety Set |
| TEAE | Treatment-emergent Adverse Event |
| VAS | Visual Analogue Scale |
| VRS | Verbal Rating Scale |

# **Definition of Terms**

| Term | Definition |
|---|---|
| Descriptive statistics | Number of subjects, mean, standard deviation, minimum, |
| | median, and maximum |
| Descriptive statistics of | Number of subjects, arithmetic mean, coefficient of |
| plasma OPA-15406 | variation, standard deviation, minimum, median, and |
| concentrations | maximum |
| Frequency distribution | Number and percentage of subjects |

#### 1 Introduction

This statistical analysis plan (SAP) documents the detailed methodology of summarization/analyses and evaluation to provide the trial data required for the preparation of a clinical study report of Trial 271-102-00002. This document has been created based on Protocol No. 271-102-00002, Version 2.0, issued on 14 Nov 2016. The pharmacokinetic analyses are detailed in Section 11.

# 2 Trial Objectives

Primary Objective: To evaluate the safety of 0.3% and 1% OPA-15406 when applied twice daily for 4 weeks in pediatric patients with atopic dermatitis (AD)

Secondary Objective: To evaluate the efficacy (dose response) and pharmacokinetics of 0.3% and 1% OPA-15406 when applied twice daily for 4 weeks in pediatric patients with AD

# 3 Trial Design

This is a multicenter, randomized, double-blind, vehicle-controlled, parallel-group comparison trial to evaluate the safety, efficacy, and pharmacokinetics of OPA-15406 ointment in pediatric patients with AD. This trial consists of the 0.3% OPA-15406 group, the 1% OPA-15406 group, and the vehicle group. The trial design is shown in Figure 3-1.

#### 1) Screening period

After obtaining written informed consent from the subject's legal guardian (if possible, after also obtaining informed assent from the subject), the investigator or subinvestigator will perform a screening examination. The period between the day of the screening examination and the end of the baseline examination is defined as the screening period (2-30 days). The subjects who meet the inclusion criteria and do not meet any of the exclusion criteria at the baseline examination will shift to the assessment period and will be dynamically allocated to the test product (0.3% or 1% formulation of OPA-15406) or the vehicle (placebo).

#### 2) Assessment period (treatment period)

For subjects meeting the inclusion criteria and not meeting any of the exclusion criteria at the baseline examination, the period between the day of the starting baseline examination and the day of the Week 4 examination (or the day of discontinuation) is defined as the assessment period. The investigational medicinal

#### Protocol 271-102-00002

product (IMP) will be administered to the treatment area from the day of the baseline examination twice daily for 4 weeks. After the baseline examination, the examination will be performed at Weeks 1, 2, and 4.

If a subject discontinues the IMP administration between the day of the baseline examination and the Week 4 examination, a withdrawal examination will be performed for that subject.

#### 3) Post-treatment observation period

The period from completion of the Week 4 examination to the day of the examination 2 weeks after the last IMP administration is defined as the post-treatment observation period. Examinations will be performed at 2 weeks after the last IMP administration. If any adverse event remained not recovered at the examination 2 weeks after the last IMP administration (or by the day of the last examination if the examination 2 weeks after the last IMP administration was not performed), it should be followed up according to the specifications.

#### 4) Trial period

The trial period for individual subjects is from the day of obtaining informed consent from the subject's legal guardian to the day of trial discontinuation or completion and does not include the follow-up period.

| | Screening period (2-30 days) | | Assessment<br>te daily adr<br>(4 wee | ministration | | Post-treatment<br>observation period<br>(2 weeks) |
|---|---|---|---|---|---|---|
| 0.3% OPA-15406 group | | <b>←</b> | | | <b>+</b> | |
| 1% OPA-15406 group | | <b>←</b> | | | <b>+</b> | |
| Vehicle group | | lack | | | <b>+</b> | |
| Informed consent | Screening examination | Start of IMP administration Baseline examination | Week 1 examination | Week 2 examination | Week 4 examination | |

: Treatment period

Figure 3-1 Trial Design Schematic

# 4 Implementation of Planned Analyses

The SAP will be finalized prior to database lock, and analyses will be performed using the final data.

# 5 Statistical Analysis Sets

# 5.1 Definitions of Analysis Sets

# 5.1.1 Efficacy Set

The efficacy set consists of all subjects who have received the IMP at least once and whose efficacy data has been obtained after the start of IMP administration.

#### 5.1.2 Safety Set

The safety set (SS) consists of all subjects who have received the IMP at least once.

# 6 Considerations for Data Analysis

#### 6.1 Software

SAS ver.9.4 (SAS Institute Inc.)

#### 6.2 Dictionaries

Coding of adverse events and medical history/complications: Medical Dictionary for Regulatory Activities (MedDRA)/J Version 20.0

Coding of prior and concomitant medications: WHO Drug Dictionary (dated 1 Mar 2016)

#### 6.3 Data Conversion and Calculation

#### 6.3.1 Response in Investigator's Global Assessment

Responders and non-responders in investigator's global assessment (IGA) are defined as follows:

- 1) Primary analysis for incidence of success in IGA
- Subjects with an IGA score of 0 (clear) or 1 (almost clear) with an improvement by at least 2 grades from baseline are defined as responders. Subjects with missing IGA data at the time of evaluation will be handled as non-responders.
- 2) Sensitivity analysis
- Subjects with an IGA score of 0 (clear) or 1 (almost clear) with an improvement by at least 2 grades from baseline are defined as responders. For subjects with missing IGA data at the time of evaluation, the last observation carried forward (LOCF) will be used.
- Subjects with an IGA score of 0 (clear) or 1 (almost clear) with an improvement by at least 2 grades from baseline are defined as responders. Observed cases (OC) will be used.

• Subjects with an improvement in IGA score to 0 (clear) or 1 (almost clear) are defined as responders. Subjects with missing IGA data at the time of evaluation will be handled as non-responders.

#### 6.3.2 Treatment Compliance

Treatment compliance = (total amount of the IMP applied from the start of administration to the assessment point<sup>1</sup>)/(sum of the specified amounts of the IMP per dose from the start of administration to the assessment point<sup>2</sup>)  $\times$  100

<sup>1</sup> [Total amount of the IMP prescribed from the start of administration to the assessment point] – [total amount of the IMP returned from the start of administration to the assessment point]

If the total amount of the IMP returned is missing, the total amount of the IMP applied from the start of administration to the assessment point will be handled as a missing value.

- <sup>2</sup> Calculation of "amount of the IMP (g) per dose"
  - 1) The subject's body surface area (BSA) (m<sup>2</sup>) will be calculated based on height and body weight at the screening examination, using the following equation.

$$BSA(m^2) = \sqrt{\frac{Ht(cm) \times Wt(kg)}{3600}}$$

2) [Amount of the IMP (g) per dose] at the assessment point will be calculated as [the subject's BSA ( $m^2$ )] × [treatment area (%) at the assessment point (including baseline)]/ $100 \times 10 \text{ g/m}^2$ .

Treatment compliance with the number of administrations will be calculated as follows:

Treatment compliance with the number of administrations = (number of administrations from the start of administration to the assessment point)/(number of days from the start of administration to the assessment point  $\times$  2)  $\times$  100

## 6.3.3 Overall Eczema Area and Severity Index Score

Overall Eczema Area and Severity Index (EASI) score is the sum of the scores for 4 body regions (face, neck, and head; upper limbs; trunk; and lower limbs). The score for each region will be calculated as shown in Table 6.3-1.

| <b>Table 6.3-1</b> | EASI Score for Each Region |
|---|---|
| Body region | Calculation of the score for each region |
| Face, neck, and head | $(E+I+Ex+L) \times score$ of affected BSA $\times$ 0.1 ( $\times$ 0.2 for children aged 2- |
| | 7 years old) |
| Upper limbs | $(E+I+Ex+L) \times score of affected BSA \times 0.2$ |
| Trunk | $(E+I+Ex+L) \times score of affected BSA \times 0.3$ |
| Lower limbs | $(E+I+Ex+L) \times score$ of affected BSA $\times$ 0.4 ( $\times$ 0.3 for children aged 2- |
| | 7 years old) |

- E = severity score of erythema; I = severity score of infiltration/papules; Ex = severity score of excoriation; L = severity score of lichenification
- Severity score: clear = 0; slight = 0.5; mild = 1; mild-moderate = 1.5; moderate = 2; severe = 2.5; very severe = 3
- Score of affected BSA (for each region): clear = 0; 1% to 9% = 1; 10% to 29% = 2; 30% to 49% = 3; 50% to 69% = 4; 70% to 89 % = 5; 90% to 100% = 6

# 6.3.4 EASI Symptom Score

Each EASI symptom score (erythema, infiltration/papules, excoriation, and lichenification) will be determined as the sum of the severity scores (Body Regions Scores) for 4 regions (face, neck, and head; upper limbs; trunk; and lower limbs) (The scores of affected BSA or multipliers will not be used in the calculation).

#### 6.4 Study Week Windows

The definitions of timepoints for analysis are described in Table 6.4-1 and Table 6.4-2. Timepoints, including unscheduled visits and visit at discontinuation, will be determined based on the number of days from the start of IMP administration. However, for Verbal Rating Scale (VRS), the timepoint will be determined based on the amount of time that has elapsed from the start of IMP administration. For efficacy variables, the data obtained between the day of the start of IMP administration and 7 days after the last IMP administration will be used in analyses. If multiple data exist within the allowable window of the timepoint, the data obtained last will be used for analyses. Data for the Last Visit will be defined as the last data obtained between the day of the start of IMP administration and 7 days after the last IMP administration (including data obtained at discontinuation) for efficacy valuables or as the last data obtained after the start of the IMP administration for safety variables.

In analyses, baseline data will be defined as data obtained on the day or at the date and time before and nearest to the start of IMP administration, including the screening data.

| Table 6.4-1 Timepoints and Allowable Windows for Efficacy Variables (Except VRS) and Safety Variables | | | | |
|---|---|---|---|---|
| Timepoint | Study Day | Allowable Window (Days After the Start of IMP Administration) | | |
| Week 1 | 8 | 1 | - | 10 |
| Week 2 | 15 | 11 | - | 21 |
| Week 4 | 29 | 22 | - | 43 |

| Table 6.4-2 Timepoints and Allowable Windows for VRS | | | |
|---|---|---|---|
| Timepoint | | low (Hou<br>Adminis | rs After the Start of stration) |
| Hour 4 | 1 | - | < 6 |
| Hour 8 | 6 | - | < 10 |
| Hour 12 | 10 | - | < 18 |
| Hour 24 | 18 | - | < 30 |
| Hour 36 | 30 | - | < 42 |
| Hour 48 | 42 | - | < 54 |
| Hour 60 | 54 | - | < 66 |
| Hour 72 | 66 | - | < 78 |
| Hour 84 | 78 | - | < 90 |
| Hour 96 | 90 | - | < 102 |
| Hour 108 | 102 | - | < 114 |
| Hour 120 | 114 | - | < 126 |
| Hour 132 | 126 | - | < 138 |
| Hour 144 | 138 | - | < 150 |
| Hour 156 | 150 | - | < 162 |
| Hour 168 | 162 | - | < 174 |

# 6.5 Handling of Missing Values

Missing data for incidence of success in IGA will be handled as described in "Section 6.3.1 Response in Investigator's Global Assessment." Other variables at each timepoint will be analyzed based on the OC and LOCF data sets.

# 6.6 Significance Level and Confidence Coefficient

No significance tests will be used in this trial; therefore, no significance levels are set. The confidence coefficient is set at two-sided 95%.

#### 6.6.1 Multiple Comparisons and Multiplicity

Multiplicity adjustment will not be conducted.

# 7 Disposition of Subjects

# 7.1 Disposition of Subjects

Data will be summarized for overall population and by age group (<7 or ≥7). The numbers of screened and randomized subjects will be provided. The following frequency distributions will be provided for overall population and by treatment group, unless otherwise specified. The frequency distribution (number and percentage relative to all subjects randomized) of subjects treated, those who completed the trial, and those who discontinued the trial will be calculated. For subjects who discontinue the trial, the frequency distribution will be calculated by reason for discontinuation.

#### 7.2 Statistical Analysis Sets

Data will be summarized for overall population and by age group (<7 or  $\ge$ 7). For the randomized subjects, the number and percentage of subjects included in the efficacy set, safety set, and pharmacokinetic analysis set will be provided.

#### 7.3 Protocol Deviations

The number and percentage of subjects with major protocol deviations will be provided for overall population and by treatment group. The number and percentage of major protocol deviations occurring in each trial site will be provided for overall population and by treatment group.

# 8 Description of Analysis Datasets

## 8.1 Demographics and Baseline Characteristics

Data will be summarized for overall population and by age group (<7 or  $\ge$ 7). For the randomized subjects, age, gender, duration of AD, body weight, height, BMI, race, baseline IGA score, and nation will be summarized for overall population and by treatment group using descriptive statistics or frequency distribution.

Affected BSA at baseline will be categorized as follows and summarized for overall population and by treatment group using frequency distribution.

Affected BSA categories:  $\geq 5\%$  to  $\leq 10\%$ ,  $\geq 10\%$  to  $\leq 30\%$ , and  $\geq 30\%$ 

#### 8.2 Medical History/Complications

Medical history and complications will be coded by MedDRA/J system organ class (SOC) and preferred term (PT). The medical history and complications will be listed, but not summarized.

#### 8.3 Prior and Concomitant Medications

For the randomized subjects, the numbers and percentages of subjects who take any concomitant medication before the start of IMP administration, during the assessment period, and after the last IMP administration will be provided by medication for the overall population and by treatment group. The medications will be coded using the WHO Drug Dictionary, and summarized by ATC Classification Level 2 and Preferred Name.

#### 8.4 Concomitant Therapies

The concomitant therapies will be listed, but not summarized.

# 9 Safety Analysis

The following safety endpoints will be analyzed in the safety set (SS).

#### 9.1 Primary Endpoint

The primary endpoint in this trial is the number and percentage of subjects experiencing adverse events (AEs). The analysis of AEs is described in Section 9.3.

# 9.2 Exposure to the IMP (Number of Subjects, Duration, and Doses)

Treatment compliance with the amount of administration and the number of administrations, calculated as described in Section 6.3.2, will be classified into the following categories, and the number and percentage of subjects will be provided for the overall population and by treatment group. The treatment compliance from baseline to Week 4 will be provided. The number and percentage of subjects who received IMP administration during each week (Week 1, Week 2, Week 3, Week 4, and every week thereafter, if necessary; Any Exposure) will be provided.

Categories of treatment compliance with the amount of administration and the number of administrations: <50%,  $\ge50\%$  to <60%,  $\ge60\%$  to <70%,  $\ge70\%$  to <80%,  $\ge80\%$  to <90%,  $\ge90\%$  to <100%,  $\ge100\%$  to <110%,  $\ge110\%$  to <120%,  $\ge120\%$ 

#### 9.3 Adverse Events

Data will be summarized for the overall population and by age group (<7 or  $\ge$ 7). All AEs will be coded using the MedDRA/J SOC and PT.

The number and percentage of subjects experiencing the following treatment-emergent adverse events (TEAEs) will be provided for the overall population and by treatment group. Skin and subcutaneous tissue disorders will also be summarized by the grade in the Common Terminology Criteria for Adverse Events (CTCAE) v4.0 Japanese JCOG edition.

- 1 TEAEs
- 2. TEAEs resulting in death
- 3. Serious TEAEs
- 4. TEAEs leading to discontinuation of IMP administration
- 5. TEAEs by severity
- 6. TEAEs by CTCAE grade (only skin and subcutaneous tissue disorders)
- 7. TEAEs at treatment areas

For TEAEs and non-serious TEAEs reported in at least 5% of subjects in any treatment group, the number and percentage of subjects will be provided for the overall population and by treatment group.

#### 9.4 Potentially Drug-related TEAEs

Potentially drug-related TEAEs (AEs for which a causal relationship with the IMP cannot be ruled out) will be summarized in the same manner as AEs. Serious potentially drug-related TEAEs will also be summarized.

#### 9.5 Clinical Laboratory Tests

For laboratory parameters (except qualitative urinalysis), measured values and changes from baseline at each timepoint will be summarized for the overall population and by treatment group using descriptive statistics. Shift tables (except qualitative urinalysis) will be created for predose and postdose values classified into normal, high, or low based on the reference range by treatment group. For qualitative urinalysis, shift tables will be created for predose and postdose values by each parameter. The number and percentage of potential Hy's Law Cases will be provided for the overall population and by treatment group. A listing of the potential Hy's Law Cases will be provided. Potential Hy's Law Cases will be defined as follows:

Potential Hy's Law Cases are defined as subjects with AST or ALT  $\geq$  3 times the upper normal limit or whose levels increase  $\geq$  3 times the initial screening value, and with an increase in total bilirubin level  $\geq$  2 times the upper normal limit or initial screening value.

#### 9.6 Vital Signs (Including Body Weight)

Measured values and changes from baseline in body weight, body temperature, blood pressure (systolic/diastolic), and pulse rate at each timepoint will be summarized for the overall population and by treatment group using descriptive statistics. For body temperature, blood pressure (systolic/diastolic), and pulse rate, the number and percentage of subjects with potentially clinically significant vital sign abnormalities (Table 16.1-1) will be computed for the overall population and by treatment group. A listing of subjects with potentially clinically significant abnormalities will be provided.

#### 9.7 Electrocardiogram (12-Lead ECG)

Measured values and changes from baseline in heart rate, PR, QRS, QT, QTc (QT interval as correlated by Bazett's formula [QTcB] and QT interval as correlated by Fridericia's formula [QTcF]), and RR intervals at each timepoint will be summarized for the overall population and by treatment group using descriptive statistics. Criteria for potentially clinically significant ECG abnormalities in heart rate, PR, QRS, QT, QTcB, and QTcF intervals will be set (Table 16.1-2), and the number and percentage of subjects who meet the criteria will be provided for the overall population and by treatment group.

# 10 Efficacy Analyses

Efficacy analyses will be performed in the efficacy set.

#### 10.1 Secondary Endpoints

#### 10.1.1 IGA

#### Incidence of success in IGA

Incidence of success in IGA at each timepoint will be compared between the 1% OPA-15406 group and the vehicle group, and between the 0.3% OPA-15406 group and the vehicle group, and p-value will be calculated, using the Cochran-Mantel-Haenszel test stratified by baseline IGA (mild or moderate). The difference in incidence of success in IGA between each OPA-15406 group and the vehicle group and its two-sided 95% confidence interval (a Mantel-Haenszel estimator of the common risk difference and its two-sided 95% confidence interval) will be computed. Additionally, two-sided 95% confidence interval for the incidence of success in IGA in each treatment group will also be calculated using Clopper-Pearson method.

The analyses will be applied to the 3 assessments defined in "Section 6.3.1 Response in Investigator's Global Assessment, 2) Sensitivity Analyses."

The SAS code to compare the incidence of success in IGA by the Cochran-Mantel-Haenszel test and to calculate the difference in incidence of success in IGA and its two-sided 95% confidence interval is shown below.

```
proc freq;
tables BaselineIGA*Treatment*Response/riskdiff(common) cmh;
run;
```

#### • Change from baseline in IGA

Based on the OC data set, the change from baseline in IGA (at Week 1, Week 2, and Week 4; if the timing of discontinuation falls within the allowable window of a timepoint, the data at discontinuation will be included as the data for the timepoint) will be analyzed using the mixed model repeated measures (MMRM) analysis with treatment (0.3% or 1% OPA-15406 group, and vehicle group), timepoint, and interaction between treatment and timepoint as factors and baseline IGA as a covariate. An unstructured covariance matrix will be used to model the within-subject errors and Kenward-Roger

method will be used to calculate the standard error of fixed-effects and the degree of freedom. If the MMRM procedure fails to converge under unstructured covariance structure, the following structure will be used in the order of 1) heterogeneous toeplitz, 2) heterogeneous autoregressive of order 1, 3) heterogeneous compound symmetry and the first (co)variance structure converging to the best fit will be used. The least square mean of each treatment group will be calculated by timepoint. The difference in the least square mean between the vehicle group and each OPA-15406 group, and the two-sided 95% confidence interval and p-value will also be calculated at Week 1, Week 2, and Week 4. The least square mean and the standard error will be plotted by timepoint for each treatment group.

The SAS code to conduct the MMRM analysis is shown below.

```
proc mixed method = reml;
  class Treatment Visit Subject;
  model Change = Treatment Visit Treatment*Visit Baseline/s ddfm = kr;
  repeated Visit/type = un sub = Subject;
  lsmeans Treatment*Visit/pdiff cl alpha = 0.05;
run;
"Baseline" represents the IGA at baseline.
```

The SAS code to use when the MMRM procedure fails to converge under the unstructured covariance structure is shown below. (Designate type = TOEPH for heterogeneous toeplitz, type = ARH(1) for heterogeneous autoregressive of order 1, and type = CSH for heterogeneous compound symmetry).

```
proc mixed method = reml empirical;
  class Treatment Visit Subject;
  model Change = Treatment Visit Treatment*Visit Baseline/s;
  repeated Visit/type= TOEPH sub = Subject;
  lsmeans Treatment*Visit/pdiff cl alpha = 0.05;
run;
```

Based on the OC and LOCF data sets, analysis of covariance (ANCOVA) model with treatment (0.3% or 1% OPA-15406 group, and vehicle group) as a factor and baseline IGA as a covariate will be applied to the change from baseline up to each timepoint. The least square mean of each treatment group will be calculated by timepoint. The difference in the least square mean between the vehicle group and each OPA-15406 group, and the two-sided 95% confidence interval and p-value will also be calculated at Week 1, Week 2, and Week 4. Based on the OC and LOCF data sets, measured values and changes from baseline in IGA at Week 1, Week 2, and Week 4 will be summarized by treatment group using descriptive statistics.

Shift tables will be created for the change from baseline in IGA  $(-3, -2, -1, \pm 0, +1, +2)$  at Week 1, Week 2, and Week 4.

# 10.1.2 Changes From Baseline in Overall EASI Score and EASI Symptom Scores

Based on the OC data set, the change from baseline in EASI score (at Week 1, Week 2, and Week 4; if the timing of discontinuation falls within the allowable window of a timepoint, the data at discontinuation will be included as the data for the timepoint) will be analyzed using the MMRM analysis with treatment (0.3% or 1% OPA-15406 group, and vehicle group), timepoint, and interaction between treatment and timepoint as factors and baseline EASI score as a covariate. An unstructured covariance matrix will be used to model the within-subject errors and Kenward-Roger method will be used to calculate the standard error of fixed-effects and the degree of freedom. If the MMRM procedure fails to converge under unstructured covariance structure, the following structure will be used in the order of 1) heterogeneous toeplitz, 2) heterogeneous autoregressive of order 1, 3) heterogeneous compound symmetry and the first (co)variance structure converging to the best fit will be used.

The least square mean of each treatment group will be calculated by timepoint. For overall EASI score, the least square mean and the standard error will be plotted by timepoint for each treatment group. The difference in the least square mean between the vehicle group and each OPA-15406 group, and the two-sided 95% confidence interval and p-value will be calculated at Week 1, Week 2, and Week 4.

Based on the OC and LOCF data sets, ANCOVA model with treatment (0.3% or 1% OPA-15406 group, and vehicle group) as a factor and baseline EASI score as a covariate will be applied to the change from baseline up to each timepoint. The least square mean in each treatment group will be calculated by timepoint. The difference in the least square

mean between the vehicle group and each OPA-15406 group, and the two-sided 95% confidence interval and p-value will be calculated at Week 1, Week 2, and Week 4. Based on the OC and LOCF data sets, measured values and changes from baseline in IGA at Week 1, Week 2, and Week 4 will be summarized by treatment group using descriptive statistics. For the overall EASI score, the mean with standard error of measured values (in the OC and LOCF data sets) will be plotted by timepoint for each treatment group.

EASI scores for body regions (face, neck, and head; upper limbs; trunk; and lower limbs) will be analyzed in the same manner as the overall EASI score.

## 10.1.3 Change From Baseline in Visual Analogue Scale for Pruritus

The change from baseline in visual analogue scale (VAS) for pruritus will be analyzed in the same manner as that in the overall EASI score or each EASI symptom score.

## 10.1.4 Change From Baseline in VRS for Pruritus up to Day 7

The change from baseline in VRS score for pruritus up to Day 7 will be analyzed in the same manner as that in overall EASI score or each EASI symptom score. Data will be collected at baseline, 4, 8, and 12 hours after the start of administration, 1 day after the start of administration (morning and night), and thereafter in the same manner up to Day 7 (morning). The same analysis will be performed by the time zone of assessment (morning or evening). Morning or evening will be determined based on the time label entered in the case report form (CRF), not using the timepoints defined in Table 6.4-2, except the baseline, which is irrespective of the time zone of assessment. Data will be collected at baseline, and the timepoints specified above on Day 1 to Day 7.

# 10.1.5 Change From Baseline in Patient-Oriented Eczema Measure Score

The change from baseline in Patient-Oriented Eczema Measure (POEM) score will be analyzed in the same manner as that in the overall EASI score or each EASI symptom score.

#### 10.1.6 Change From Baseline in Overall Percentage Affected BSA

The change from baseline in overall percentage affected BSA will be analyzed in the same manner as that in the overall EASI score or each EASI symptom score.

# 10.1.7 Percent Changes From Baseline in Overall EASI Score, EASI Symptom Scores, VAS for Pruritus, and POEM Scores

The percent changes from baseline in overall EASI score, EASI symptom scores, EASI scores for body regions, VAS for pruritus, and POEM score will be analyzed in the same manner as the changes from baseline in the respective scores.

#### 10.1.8 Time to Response in IGA

For the time to response in IGA (days to the first response in IGA in each subject), a cumulative response rate will be computed by treatment group using the Kaplan-Meier method and plotted. At each timepoint, the number of subjects (at risk), the p-value of the log-rank test comparing the vehicle group and each OPA-15406 group, and the time until one half of the subjects have achieved a response (medial survival time [MST]) will be provided. Subjects with an IGA of 0 (clear) or 1 (almost clear) with an improvement by at least 2 grades from the baseline are defined as responders. The starting point is the baseline. Subjects who have failed to achieve a response will be treated as censored on the day of the final IGA assessment.

#### 10.1.9 Time to Response in VRS

The time to response in VRS (time to the first response in VRS in each subject) will be analyzed in the same manner as the time to response in IGA. Subjects with a VRS score of 0 (none) or 1 (mild) with an improvement by at least 1 grade from the baseline are defined as responders. The starting point is baseline. Subjects who have failed to achieve a response will be treated as censored on the day of the final VRS assessment.

#### 10.2 Other Efficacy Endpoints

Not applicable.

#### 10.3 Adjustments for Covariates

In the analysis of the incidence of success in IGA, the Cochran-Mantel-Haenszel test stratified by baseline IGA (mild or moderate) will be conducted.

#### 10.4 Subgroup Analysis

Incidence of success in IGA will also be analyzed in the following subgroups in the same manner as described in Section 10.1.1.

Age: <7 or  $\ge 7$  years old

Gender: Male or female

Baseline IGA score: 2 (mild) or 3 (moderate)

# 11 Pharmacokinetic Analyses

# 11.1 Pharmacokinetics Analysis Set

The pharmacokinetic analysis set consists of all subjects who have received the IMP at least once and have at least one evaluable plasma drug concentration measured.

#### 11.2 Pharmacokinetic Endpoints

• Plasma trough concentration of OPA-15406 (predose at Week 1 and Week 4)

#### 11.3 Method of Calculation of Pharmacokinetic Endpoints

- 1) Plasma concentrations below the lower limit of quantification will be treated as zero (ng/mL) for the calculation of descriptive statistics.
- 2) Plasma trough concentrations will be handled as follows:
- If the time of the blood sampling was within 6 hours from the last IMP administration, the sampling point will be excluded from the analysis.
- If the treatment area (%) was changed (including non-compliance of IMP) within 3 days before the sampling point, the sampling point will be excluded from the analysis.
- 3) The timepoint of blood sampling for the pharmacokinetic endpoint at withdrawal will be handled as follows: If the blood sampling at withdrawal meets neither of the exclusion criteria in (2) and falls within the allowable window shown below, the sampling point will be included in the analyses. If the blood sampling at

withdrawal coincides with any pharmacokinetic timepoint, the blood sampling at withdrawal will not be included in the analyses.

| Timepoint | Study Day | Allowable | Windo | w (Day) |
|-----------|-----------|-----------|-------|---------|
| Baseline | 1 | | - | 1 |
| Week 1 | 8 | 4 | - | 22 |
| Week 4 | 29 | 23 | - | 50 |

4) The dose used for the dose adjustment of concentration will be calculated as follows:

#### 11.4 Method of Display

- 1) When plotting the plasma drug concentration-time profile, arithmetic means and standard deviations will be used.
- 2) Descriptive statistics of the plasma trough concentrations and dose(mg)-normalized plasma trough concentrations will be calculated by treatment group and pharmacokinetic timepoint.
- 3) Descriptive statistics of the total treatment area (%) will be calculated by treatment group and pharmacokinetic timepoint.
- 4) In 2) or 3) above, when the number of analyzed subjects is zero (0), only the number of subjects will be calculated; when only one (1) subject is analyzed, only the number of subjects, arithmetic mean, and geometric mean will be calculated; and when two (2) subjects are analyzed, only the number of subjects, arithmetic mean, geometric mean, and maximum and minimum values will be calculated.

#### 11.5 Handling of Values

Among descriptive statistics, the number of subjects will be displayed in integers, and minimum and maximum will be displayed as it is in the same number of digits (n-digit) as that of an individual value of the target data. For arithmetic mean, geometric mean, median, and standard deviation values, a value of "n + 1" figures will be rounded off to obtain a value of "n" figures so that the number of digits will be the same number of digits (n-digit) as that of an individual value of the target data. For coefficient of variation, 2 decimal places will be rounded to obtain 1 decimal place.

# 12 Rationale for Target Number of Subjects

# 12.1 Target Number of Subjects

60 subjects

#### 12.2 Rationale for the Number of Subjects

The sample size of 20 subjects for each group, a total of 60 subjects, has been established in consideration of the feasibility of the trial and the number of subjects needed to evaluate efficacy and safety. Assuming that the probabilities of success in IGA for each group are the same as those in the phase 2 trial outside Japan (271-12-205), the expected incidence of success in the 1% OPA-15406 group, the 0.3% OPA-15406 group, and the vehicle group is 20.93%, 14.63%, and 2.7%, respectively. In that case, the probability of the 1% group > the vehicle group, the 0.3% group > the vehicle group, and the 1% group minus the vehicle group > 10% in the point estimate of incidence of success is 96.2%, 88.3%, and 71.5%, respectively. Also, the probability of the 1% group > the 0.3% group > the vehicle group in point estimate of incidence of success is 60.6%.

# 13 Changes From Analysis Planned in the Protocol

#### 13.1 Changes From the Efficacy Analyses Planned in the Protocol

• The factors/covariates included in the MMRM or ANCOVA model were described consistently. A categorical variable included in the model was described as a factor, and a continuous variable as a covariate.

Rationale for change: To further clarify the analytical methods

# 13.2 Changes From the Pharmacokinetic Analyses Planned in the Protocol

- The descriptive statistics of the plasma trough concentrations of OPA-15406 will not be calculated by affected BSA at baseline. The plasma trough concentrations of OPA-15406 will be normalized by dose (mg), not by affected BSA.
   Rationale for change: Calculation of dose-normalized plasma trough concentration was considered adequate, the concentrations will not be computed by or normalized by affected BSA.
- The descriptive statistics for age, treatment area at baseline, and amount of administration will not be calculated by the affected BSA.

Protocol 271-102-00002

Rationale for change: These were considered not necessary for interpretation of the data.

• The descriptive statistics of total treatment area (%) will be calculated by treatment group and pharmacokinetic timepoint.

Rationale for change: These were considered necessary for interpretation of the data.

# 14 References

Not applicable.

# 15 Revision History

Not applicable.

| Table 15-1 Revision History | | | | | |
|---|---|---|---|---|---|
| Version Number | Date of Revision | Section | Original Description | Revised Description | Reason for Revision |
| _ | _ | _ | _ | _ | _ |

# 16 Appendix

# 16.1 Criteria for Potentially Clinically Significant

| Table 16.1-1 Criteria for Potentially Clinically Significant Vital Sign Abnormalities | | |
|---|---|---|
| TEST | CRITERIA 1 | CRITERIA 2 |
| DIASTOLIC BLOOD | DIASTOLIC BLOOD PRESSURE | DIASTOLIC BLOOD PRESSURE |
| PRESSURE (MMHG) | (mmHg) < 50 AND DECREASE >= | (mmHg) > 105 AND INCREASE |
| | 15 | >= 15 |
| HEART RATE | HEART RATE (BPM) < 50 AND | HEART RATE (BPM) > 120 AND |
| (BEATS/MIN) | DECREASE >= 15 | INCREASE >= 15 |
| SYSTOLIC BLOOD | SYSTOLIC BLOOD PRESSURE | SYSTOLIC BLOOD PRESSURE |
| PRESSURE (MMHG) | (mmHg) < 90 AND DECREASE >= | (mmHg) > 180 AND INCREASE |
| | 20 | >= 20 |
| TEMPERATURE (°C) | - | TEMPERATURE (°C) $\geq$ 37.8 |
| , í | | AND INCREASE $\geq 1.1$ °C |
| WEIGHT (KG) | WEIGHT (kg) DECREASE >= 7% | WEIGHT (kg) INCREASE >= 7% |

| <b>Table 16.1-2</b> | Criteria for Potentially Clinically Significant ECG | |
|---|---|---|
| | Abnormalities | |
| CLASSIFICATION | CATEGORY | CRITERIA |
| VENT RATE | NOTABLE | 25% INCREASE FROM BASELINE AND |
| OUTLIERS | INCREASES | VENTRICULAR RATE > 100 BPM |
| VENT RATE | NOTABLE | 25% DECREASE FROM BASELINE AND |
| OUTLIERS | DECREASES | VENTRICULAR RATE < 50 BPM |
| PR OUTLIERS | NOTABLE CHANGES | >= 25% CHANGE FROM BASELINE WHEN PR > |
| | | 200 MSEC |
| QRS OUTLIERS | NOTABLE CHANGES | >= 25% CHANGE FROM BASELINE WHEN QRS |
| | | > 100 MSEC |
| QT | NEW ONSET (>= 450 | NEW ONSET (>= 450 MSEC) IN QT MEANS A |
| | MSEC) | SUBJECT WHO ATTAINS A VALUE >= 450 |
| | | MSEC DURING TREATMENT PERIOD BUT |
| | | NOT AT EACH BASELINE |
| QTcB | NEW ONSET (>= 450 | NEW ONSET (>= 450 MSEC IN MALE OR >= 470 |
| | MSEC) IN MALE OR | MSEC IN FEMALE) IN QTCB MEANS A |
| | (>= 470 MSEC) IN | SUBJECT WHO ATTAINS A VALUE >= 450 OR |
| | FEMALE | >= 470 MSEC DURING TREATMENT PERIOD |
| | | BUT NOT AT EACH BASELINE |
| QTcB | NEW ONSET (>= 450 | NEW ONSET (>= 450 MSEC) AND >= 10% |
| | MSEC) AND $\geq 10\%$ | INCREASE IN QTCB MEANS A SUBJECT WHO |
| | INCREASE | ATTAINS A VALUE >= 450 MSEC AND >= 10% |
| | | INCREASE DURING TREATMENT PERIOD |
| | | BUT NOT AT EACH BASELINE |
| QTcB | INCREASE 30 - 60 | INCREASE IN CHANGE FROM BASELINE |
| | MSEC | VALUE >= 30 AND <= 60 MSEC |
| QTcB | INCREASE > 60 MSEC | INCREASE IN CHANGE FROM BASELINE |
| | | VALUE > 60 MSEC |

| Table 16.1-2 | Criteria for Potentially Clinically Significant ECG<br>Abnormalities | |
|---|---|---|
| CLASSIFICATION | CATEGORY | CRITERIA |
| QTcF | NEW ONSET (>= 450 | NEW ONSET (>= 450 MSEC IN MALE OR >= 470 |
| | MSEC) IN MALE OR | MSEC IN FEMALE) IN QTCB MEANS A |
| | (>= 470 MSEC) IN | SUBJECT WHO ATTAINS A VALUE >= 450 OR |
| | FEMALE | >= 470 MSEC DURING TREATMENT PERIOD |
| | | BUT NOT AT EACH BASELINE |
| QTcF | NEW ONSET (>= 450 | NEW ONSET (>= 450 MSEC) AND >= 10% |
| | MSEC) AND $\geq 10\%$ | INCREASE IN QTCB MEANS A SUBJECT WHO |
| | INCREASE | ATTAINS A VALUE >= 450 MSEC AND >= 10% |
| | | INCREASE DURING TREATMENT PERIOD |
| | | BUT NOT AT EACH BASELINE |
| QTcF | INCREASE 30 - 60 | INCREASE IN CHANGE FROM BASELINE |
| | MSEC | $VALUE >= 30 AND \le 60 MSEC$ |
| QTcF | INCREASE > 60 MSEC | INCREASE IN CHANGE FROM BASELINE |
| | | VALUE > 60 MSEC |

#### 16.2 Table of Contents

- CT-1 Subject Disposition
- CT-2 Reasons for Discontinuation
- CT-3 Demographic Characteristics
- CT-4.1 Concomitant Medications: Medications Taken Prior to Start of Study Therapy
- CT-4.2 Concomitant Medications: Medications Taken During Study Therapy
- CT-4.3 Concomitant Medications: Medications Taken After Study Therapy
- CT-5.1.1 Analysis of Responder Rate for Overall IGA Score
- CT-5.1.2 Sensitivity Analysis of Responder Rate for Overall IGA Score LOCF
- CT-5.1.3 Sensitivity Analysis of Responder Rate for Overall IGA Score OC
- CT-5.1.4 Sensitivity Analysis of Responder Rate for Overall IGA Score Revised Responder Definition
- CT-5.1.5 Shift Tables of Overall IGA Score OC
- CT-5.1.6 Shift Tables of Overall IGA Score LOCF
- CT-5.2.1 Analysis of Baseline and Change from Baseline in Overall IGA Score MMRM
- CT-5.2.2 Analysis of Baseline and Change from Baseline in Overall IGA Score ANCOVA OC

- CT-5.2.3 Analysis of Baseline and Change from Baseline in Overall IGA Score ANCOVA LOCF
- CT-5.3.1.1 Analysis of Baseline and Change from Baseline in Overall EASI Score MMRM
- CT-5.3.1.2 Analysis of Baseline and Change from Baseline in Overall EASI Score ANCOVA OC
- CT-5.3.1.3 Analysis of Baseline and Change from Baseline in Overall EASI Score ANCOVA LOCF
- CT-5.3.1.4 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score MMRM
- CT-5.3.1.5 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score ANCOVA OC
- CT-5.3.1.6 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score ANCOVA LOCF
- CT-5.3.2.1 Analysis of Baseline and Change from Baseline in Overall EASI Score, Erythema MMRM
- CT-5.3.2.2 Analysis of Baseline and Change from Baseline in Overall EASI Score, Erythema ANCOVA OC
- CT-5.3.2.3 Analysis of Baseline and Change from Baseline in Overall EASI Score, Erythema ANCOVA LOCF
- CT-5.3.2.4 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Erythema MMRM
- CT-5.3.2.5 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Erythema ANCOVA OC
- CT-5.3.2.6 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Erythema ANCOVA LOCF
- CT-5.3.3.1 Analysis of Baseline and Change from Baseline in Overall EASI Score, Induration/Papulation MMRM
- CT-5.3.3.2 Analysis of Baseline and Change from Baseline in Overall EASI Score, Induration/Papulation ANCOVA OC
- CT-5.3.3.3 Analysis of Baseline and Change from Baseline in Overall EASI Score, Induration/Papulation ANCOVA LOCF

- CT-5.3.3.4 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Induration/Papulation MMRM
- CT-5.3.3.5 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Induration/Papulation ANCOVA OC
- CT-5.3.3.6 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Induration/Papulation ANCOVA LOCF
- CT-5.3.4.1 Analysis of Baseline and Change from Baseline in Overall EASI Score, Excoriation MMRM
- CT-5.3.4.2 Analysis of Baseline and Change from Baseline in Overall EASI Score, Excoriation ANCOVA OC
- CT-5.3.4.3 Analysis of Baseline and Change from Baseline in Overall EASI Score, Excoriation ANCOVA LOCF
- CT-5.3.4.4 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Excoriation MMRM
- CT-5.3.4.5 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Excoriation ANCOVA OC
- CT-5.3.4.6 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Excoriation ANCOVA LOCF
- CT-5.3.5.1 Analysis of Baseline and Change from Baseline in Overall EASI Score, Lichenification MMRM
- CT-5.3.5.2 Analysis of Baseline and Change from Baseline in Overall EASI Score, Lichenification ANCOVA OC
- CT-5.3.5.3 Analysis of Baseline and Change from Baseline in Overall EASI Score, Lichenification ANCOVA LOCF
- CT-5.3.5.4 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Lichenification MMRM
- CT-5.3.5.5 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Lichenification ANCOVA OC
- CT-5.3.5.6 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, Lichenification ANCOVA LOCF
- CT-5.3.6.1 Analysis of Baseline and Change from Baseline in Overall EASI Score, HEAD/NECK MMRM

- CT-5.3.6.2 Analysis of Baseline and Change from Baseline in Overall EASI Score, HEAD/NECK ANCOVA OC
- CT-5.3.6.3 Analysis of Baseline and Change from Baseline in Overall EASI Score, HEAD/NECK ANCOVA LOCF
- CT-5.3.6.4 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, HEAD/NECK MMRM
- CT-5.3.6.5 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, HEAD/NECK ANCOVA OC
- CT-5.3.6.6 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, HEAD/NECK ANCOVA LOCF
- CT-5.3.7.1 Analysis of Baseline and Change from Baseline in Overall EASI Score, UPPER LIMBS MMRM
- CT-5.3.7.2 Analysis of Baseline and Change from Baseline in Overall EASI Score, UPPER LIMBS ANCOVA OC
- CT-5.3.7.3 Analysis of Baseline and Change from Baseline in Overall EASI Score, UPPER LIMBS ANCOVA LOCF
- CT-5.3.7.4 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, UPPER LIMBS MMRM
- CT-5.3.7.5 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, UPPER LIMBS ANCOVA OC
- CT-5.3.7.6 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, UPPER LIMBS ANCOVA LOCF
- CT-5.3.8.1 Analysis of Baseline and Change from Baseline in Overall EASI Score, TRUNK MMRM
- CT-5.3.8.2 Analysis of Baseline and Change from Baseline in Overall EASI Score, TRUNK ANCOVA OC
- CT-5.3.8.3 Analysis of Baseline and Change from Baseline in Overall EASI Score, TRUNK ANCOVA LOCF
- CT-5.3.8.4 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, TRUNK MMRM
- CT-5.3.8.5 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, TRUNK ANCOVA OC

- CT-5.3.8.6 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, TRUNK ANCOVA LOCF
- CT-5.3.9.1 Analysis of Baseline and Change from Baseline in Overall EASI Score, LOWER LIMBS MMRM
- CT-5.3.9.2 Analysis of Baseline and Change from Baseline in Overall EASI Score, LOWER LIMBS ANCOVA OC
- CT-5.3.9.3 Analysis of Baseline and Change from Baseline in Overall EASI Score, LOWER LIMBS ANCOVA LOCF
- CT-5.3.9.4 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, LOWER LIMBS MMRM
- CT-5.3.9.5 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, LOWER LIMBS ANCOVA OC
- CT-5.3.9.6 Analysis of Baseline and Percent Change from Baseline in Overall EASI Score, LOWER LIMBS ANCOVA LOCF
- CT-5.4.1 Analysis of Baseline and Change from Baseline in VAS for Pruritus Score MMRM
- CT-5.4.2 Analysis of Baseline and Change from Baseline in VAS for Pruritus Score ANCOVA OC
- CT-5.4.3 Analysis of Baseline and Change from Baseline in VAS for Pruritus Score ANCOVA LOCF
- CT-5.4.4 Analysis of Baseline and Percent Change from Baseline in VAS for Pruritus Score MMRM
- CT-5.4.5 Analysis of Baseline and Percent Change from Baseline in VAS for Pruritus Score ANCOVA OC
- CT-5.4.6 Analysis of Baseline and Percent Change from Baseline in VAS for Pruritus Score ANCOVA LOCF
- CT-5.5.1 Analysis of Baseline and Change from Baseline in Overall Percentage Affected Body Surface Area MMRM
- CT-5.5.2 Analysis of Baseline and Change from Baseline in Overall Percentage Affected Body Surface Area ANCOVA OC
- CT-5.5.3 Analysis of Baseline and Change from Baseline in Overall Percentage Affected Body Surface Area ANCOVA LOCF

- CT-5.6.1 Analysis of Baseline and Change from Baseline in POEM Score MMRM
- CT-5.6.2 Analysis of Baseline and Change from Baseline in POEM Score ANCOVA OC
- CT-5.6.3 Analysis of Baseline and Change from Baseline in POEM Score ANCOVA LOCF
- CT-5.6.4 Analysis of Baseline and Percent Change from Baseline in POEM Score MMRM
- CT-5.6.5 Analysis of Baseline and Percent Change from Baseline in POEM Score ANCOVA OC
- CT-5.6.6 Analysis of Baseline and Percent Change from Baseline in POEM Score ANCOVA LOCF
- CT-5.7.1 Analysis of Baseline and Change from Baseline in VRS for Pruritus Score MMRM
- CT-5.7.2 Analysis of Baseline and Change from Baseline in VRS for Pruritus Score ANCOVA OC
- CT-5.7.3 Analysis of Baseline and Change from Baseline in VRS for Pruritus Score ANCOVA LOCF
- CT-5.7.4 Analysis of Baseline and Change from Baseline in VRS for Pruritus Score (Morning / Evening) MMRM
- CT-5.7.5 Analysis of Baseline and Change from Baseline in VRS for Pruritus Score (Morning / Evening) ANCOVA OC
- CT-5.8.1 Subgroup Analysis of Responder Rate for Overall IGA Score by Age
- CT-5.8.2 Subgroup Analysis of Responder Rate for Overall IGA Score by Gender
- CT-5.8.3 Subgroup Analysis of Responder Rate for Overall IGA Score by IGA Score at Baseline
- CT-7.1.1 Summary of Treatment Compliance
- CT-7.1.2 Summary of Treatment Compliance for Number of Administrations
- CT-7.2 Extent of Exposure to Trial Medication
- CT-8.1.1 Adverse Events (All Causalities)
- CT-8.1.2 Adverse Events According to Application Site (All Causalities)
- CT-8.2.1.1 Incidence of Treatment-emergent Adverse Events by System Organ Class

- CT-8.2.1.2 Incidence of Treatment-emergent Adverse Events by System Organ Class
- CT-8.2.1.3 Incidence of Treatment-emergent Adverse Events by System Organ Class
- CT-8.2.2.1 Incidence of Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.2.2.2 Incidence of Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.2.2.3 Incidence of Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.2.3.1 Incidence of Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity
- CT-8.2.3.2 Incidence of Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity
- CT-8.2.3.3 Incidence of Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity
- CT-8.2.4.1 Incidence of Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade
- CT-8.2.4.2 Incidence of Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade
- CT-8.2.4.3 Incidence of Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade
- CT-8.3.1.1 Incidence of Potentially Drug-Related Treatment-emergent Adverse Events by System Organ Class
- CT-8.3.1.2 Incidence of Potentially Drug-Related Treatment-emergent Adverse Events by System Organ Class
- CT-8.3.1.3 Incidence of Potentially Drug-Related Treatment-emergent Adverse Events by System Organ Class
- CT-8.3.2.1 Incidence of Potentially Drug-Related Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.3.2.2 Incidence of Potentially Drug-Related Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.3.2.3 Incidence of Potentially Drug-Related Treatment-emergent Adverse Events by System Organ Class and Preferred Term

- CT-8.3.3.1 Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity
- CT-8.3.3.2 Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity
- CT-8.3.3.3 Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity
- CT-8.3.4.1 Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade
- CT-8.3.4.2 Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade
- CT-8.3.4.3 Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade
- CT-8.4.1.1 Incidence of Deaths due to Treatment-emergent Adverse Events by System Organ Class
- CT-8.4.1.2 Incidence of Deaths due to Treatment-emergent Adverse Events by System Organ Class
- CT-8.4.1.3 Incidence of Deaths due to Treatment-emergent Adverse Events by System Organ Class
- CT-8.4.2.1 Incidence of Deaths due to Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.4.2.2 Incidence of Deaths due to Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.4.2.3 Incidence of Deaths due to Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.5.1.1 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class
- CT-8.5.1.2 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class
- CT-8.5.1.3 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class
- CT-8.5.2.1 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term

- CT-8.5.2.2 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.5.2.3 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term
- CT-8.5.3.1 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity
- CT-8.5.3.2 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity
- CT-8.5.3.3 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Severity
- CT-8.5.4.1 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade
- CT-8.5.4.2 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade
- CT-8.5.4.3 Incidence of Serious Treatment-emergent Adverse Events by System Organ Class, Preferred Term and CTCAE Grade
- CT-8.6.1.1 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class
- CT-8.6.1.2 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class
- CT-8.6.1.3 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class
- CT-8.6.2.1 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class and Preferred Term
- CT-8.6.2.2 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class and Preferred Term
- CT-8.6.2.3 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class and Preferred Term
- CT-8.6.3.1 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class and Preferred Term
- CT-8.6.3.2 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class and Preferred Term

- CT-8.6.3.3 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class and Preferred Term
- CT-8.6.4.1 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class and Preferred Term
- CT-8.6.4.2 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class and Preferred Term
- CT-8.6.4.3 Incidence of Treatment-emergent Adverse Events Resulting in Discontinuation from Study by System Organ Class and Preferred Term
- CT-8.7.1.1 Incidence of Treatment-emergent Adverse Events Greater Than or Equal to 5% in Any Group by System Organ Class and Preferred Term
- CT-8.7.1.2 Incidence of Treatment-emergent Adverse Events Greater Than or Equal to 5% in Any Group by System Organ Class and Preferred Term
- CT-8.7.1.3 Incidence of Treatment-emergent Adverse Events Greater Than or Equal to 5% in Any Group by System Organ Class and Preferred Term
- CT-8.8.1.1 Incidence of Non-Serious Treatment-emergent Adverse Events Greater Than or Equal to 5% in Any Group by System Organ Class and Preferred Term
- CT-8.8.1.2 Incidence of Non-Serious Treatment-emergent Adverse Events Greater Than or Equal to 5% in Any Group by System Organ Class and Preferred Term
- CT-8.8.1.3 Incidence of Non-Serious Treatment-emergent Adverse Events Greater Than or Equal to 5% in Any Group by System Organ Class and Preferred Term
- CT-8.9.1.1 Incidence of Treatment-emergent Adverse Events by System Organ Class and Preferred Term According to Application Site
- CT-8.9.1.2 Incidence of Treatment-emergent Adverse Events by System Organ Class and Preferred Term According to Application Site
- CT-8.9.1.3 Incidence of Treatment-emergent Adverse Events by System Organ Class and Preferred Term According to Application Site
- CT-8.10.1.1 Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class and Preferred Term According to Application Site
- CT-8.10.1.2 Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class and Preferred Term According to Application Site
- CT-8.10.1.3 Incidence of Potentially Drug-related Treatment-emergent Adverse Events by System Organ Class and Preferred Term According to Application Site

- CT-9.1 Listing of Deaths
- CT-9.2 Listing of Serious Adverse Events
- CT-9.3 Listing of Study Drug Discontinuations Due to Adverse Events
- CT-9.4 Incidence of Potential Hy's Law Cases
- CT-9.5 Listing of Potential Hy's Law Cases by Subject
- CT-10.1.1 Mean Change From Baseline in Laboratory Test Values: Serum Chemistry
- CT-10.1.2 Mean Change From Baseline in Laboratory Test Values: Hematology
- CT-10.2.1 Shift Tables of Clinical Laboratory Test Results: Serum Chemistry
- CT-10.2.2 Shift Tables of Clinical Laboratory Test Results: Hematology
- CT-10.2.3 Shift Tables of Clinical Laboratory Test Results: Urinalysis
- CT-11.1 Mean Change From Baseline in Vital Sign Parameters
- CT-11.2 Listing of Vital Signs Abnormalities
- CT-11.3 Incidence of Potential Clinical Significance in Vital Signs
- CT-11.4 Criteria for Vital Signs Potential Clinical Significance
- CT-12.1 Mean Change From Baseline in ECG Evaluations
- CT-12.2 Incidence of Categorical Changes in ECG Evaluations
- CT-12.3 Listing of Categorical Changes in ECG Evaluations
- CT-12.4 Criteria for Categorical Changes in ECG Evaluations
- PKT-1.1 Individual and Summary of OPA-15406 Plasma Trough Concentrations Following Topical Administration of 0.3 % OPA-15406 Ointment to Child Subjects With Atopic Dermatitis
- PKT-1.2 Individual and Summary of OPA-15406 Plasma Trough Concentrations Following Topical Administration of 1 % OPA-15406 Ointment to Child Subjects With Atopic Dermatitis
- PKT-2.1 Individual and Summary of Normalized OPA-15406 Plasma Trough Concentrations by Dose Derived From % BSA Treated Following Topical Administration of 0.3 % OPA-15406 Ointment to Child Subjects With Atopic Dermatitis

#### Protocol 271-102-00002

PKT-2.2 Individual and Summary of Normalized OPA-15406 Plasma Trough Concentrations by Dose Derived From % BSA Treated Following Topical Administration of 1 % OPA-15406 Ointment to Child Subjects With Atopic Dermatitis

PKF-1.1 Mean OPA-15406 Plasma Trough Concentrations Following Topical Administration of OPA-15406 Ointment to Child Subject With Atopic Dermatitis

PKF-1.2 Mean Normalized OPA-15406 Plasma Trough Concentrations by Dose Derived From % BSA Treated Following Topical Administration of OPA-15406 Ointment to Child Subject With Atopic Dermatitis

PDATA-1.1 Inclusion and Exclusion Criteria

PDATA-1.2 Subject Disposition

PDATA-2.1 Medical History

PDATA-2.2 History of Atopic Dermatitis

PDATA-3.1 Concomitant Medications: Medications Taken Prior to Start of Study Therapy

PDATA-3.2 Concomitant Medications: Medications Taken During Study Therapy

PDATA-3.3 Concomitant Medications: Medications Taken After Study Therapy

PDATA-4.1 Exposure to Trial Medication

PDATA-4.2 Listing of Trial Medication by Subject

PDATA-5.1 Physical Examination

PDATA-6 Adverse Events

PDATA-7 Vital Signs

PDATA-8 Electrocardiogram Results

PDATA-9 Blood Sampling for Pharmacokinetics

PDATA-10 Screening Failures

PDATA-11 Protocol Deviations (Major) - CRF

PDATA-12 Patch Application and Removal

PDATA-13 Eczema Area and Severity Index

PDATA-14 Visual Analog Scale for Pruritus

| Protocol | 271 | -10 | 12-0 | 0000 | 2 |
|----------|-----|-------|------|------|---|
| TIOROGOT | 21 | - 1 ( | 12-1 | ハハハ | 1 |

PDATA-15 Verbal Rating Scale

PDATA-16 Overall Investigator's Global Assessment of Disease Severity

PDATA-17 Patient-Oriented Eczema Measure

PDATA-18 Affected Body Surface Area

PDATA-19 Treatment Area

DREAS-1 Discontinued Subjects and Reasons for Discontinuations

DEMOG-1 Demographic Characteristics

**DEMOG-2 Informed Consent** 

AE-1 Adverse Events

SMED-1 Investigational Medicinal Product Compliance

SMED-2 Actual Exposure to Study Medication

SMED-3 Investigational Medicinal Product Compliance for Number of Administrations

EFF-1 Change from Baseline in IGA Score and Response with Overall IGA Score

EFF-2 Change from Baseline in Total EASI Score

EFF-3 Change from Baseline in EASI Score, Erythema

EFF-4 Change from Baseline in EASI Score, Induration/Papulation

EFF-5 Change from Baseline in EASI Score, Excoriation

EFF-6 Change from Baseline in EASI Score, Lichenification

EFF-7 Change from Baseline in EASI Score, HEAD/NECK

EFF-8 Change from Baseline in EASI Score, UPPER LIMBS

EFF-9 Change from Baseline in EASI Score, TRUNK

EFF-10 Change from Baseline in EASI Score, LOWER LIMBS

#### Protocol 271-102-00002

- EFF-11 Change from Baseline in VAS Score
- EFF-12 Change from Baseline in Overall Percentage Affected Body Surface Area
- EFF-13 Change from Baseline in POEM Score
- EFF-14 Change from Baseline in VRS Score
- LAB-1 Laboratory Test Results: Serum Chemistry
- LAB-2 Laboratory Test Results: Hematology
- LAB-3 Laboratory Test Results: Urinalysis
- PDEV-1 Summary of Subjects with Major Protocol Deviations by Type of Deviation
- SUBEX-1 Subjects Excluded From Analysis Set